CLINICAL TRIAL: NCT03999528
Title: 14-3-3η Protein, Disease Activity and Bone Mineral Density, in Female Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abogamal, Professor, Al-Azhar University
Other Study IDs: Rheu-med.9med.research
Record Dates: First submitted 2019-06-10; First posted 2019-06-26 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis; Osteoporosis
Keywords: 14-3-3η Protein
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: RA Patients
  Interventions: Diagnostic Test: 14-3-3η Protein assay
- control group: normal control
  Interventions: Diagnostic Test: 14-3-3η Protein assay

INTERVENTIONS:
Diagnostic Test: 14-3-3η Protein assay — blood sampling for assessment of serum 14-3-3η Protein

SUMMARY:
Is to investigate the relation between 14-3-3η protein, disease activity, and bone mineral density in female patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Methods: all patients in the study will subject to:

* Clinical assessment, WT, Height ,BMI, parity, medications,
* DAS 28.
* Serum 14-3-3η protein.
* DEXA scan.

Grouping:

* Group I: RA Patients with low BMD.
* Group II: RA Patients with normal BMD.
* Group III: normal control.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis according to ACR 2010 criteria with at least one year duration.
* Premenopausal females.
* On conventional DMARD with maximum 5 mg steroids.

Exclusion Criteria:

* Biological treatment.
* Previous antiresorptive treatment, or bone anabolics.
* High dose corticosteroid.
* Chronic renal or kidney disease.
* Medications affecting bone metabolism.
* Thyroid or adrenal dysfunction,

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with rheumatoid arthritis attending the Rheumatology department, at Al-Azhar faculty of medicine from May 2019 to August 2019
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
14-3-3η Protein and RA disease activity | three months
  percent of active RA disease and study the correlation between 14-3-3η Protein and RA disease activity

SECONDARY OUTCOMES:
14-3-3η Protein and osteoporosis in RA patients | three months
  percent of low BMD and study the correlation between 14-3-3η Protein and osteoporosis in RA patients

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ABOGAMAL, Study Chair — Al-Azhar Faculty of medicine- Cairo
Locations (1):
- Al-Azhar Faculty of medicine, Rheumatology Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No